CLINICAL TRIAL: NCT05110599
Title: Bryophyllum Pinnatum Treatment of Anxiety Related to Signs of Preterm Birth: a Randomised, Double-blind, Placebo-controlled Study as Investigator-Initiated Trial
Brief Title: Bryophyllum Pinnatum Treatment of Anxiety Related to Signs of Preterm Birth
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment and expired study medication.
Sponsor: Christian Haslinger (Other)
Responsible Party: Sponsor-Investigator, Christian Haslinger, Principal Investigator, University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BASEC-Nr. 2021-00941
Record Dates: First submitted 2021-10-05; First posted 2021-11-08 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Preterm Labor; Anxiety
Keywords: Bryophyllum pinnatum; Anxiety; Preterm labor; Sleep quality; Phytotherapy
MeSH Terms: conditions — Obstetric Labor, Premature; Anxiety Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: 48 h after hospitalisation patients can be randomized to the Bryophyllum group or the placebo group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bryophyllum 50% (Active Comparator): Participants of the verum group take Bryophyllum 50% chewable tablets starting the day after study inclusion. Participants take 2 tablets, four times a day for 2 weeks. If the birth takes place before the end of the 2 weeks, the study participation is terminated early.
  Interventions: Drug: Bryophyllum 50% chewable tablets
- Placebo (Placebo Comparator): Participants of the control group take Placebo chewable tablets starting the day after study inclusion. Participants take 2 tablets, four times a day for 2 weeks. If the birth takes place before the end of the 2 weeks, the study participation is terminated early.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bryophyllum 50% chewable tablets — Each 350 mg tablet corresponds to 170 mg of leave press juice from Bryophyllum pinnatum, dried down to 17 mg by mixing with lactose; 100 mg dried BP matter in 1 g
  Arms: Bryophyllum 50%
Other: Placebo — Lactose with adaption in appearance and tast
  Arms: Placebo

SUMMARY:
The present IIT (Investigator-Initiated Trial) study is a prospective, randomised, placebo-controlled, double blind trial.

Women hospitalised with signs of preterm birth can be recruited for the study. Participants will take study medication for 2 weeks (or until birth) and fill out a questionnaire at 3 time points (at baseline, after 1 week and after 2 weeks) to assess state of anxiety and sleep quality. Furthermore, information regarding adverse events and the further course of the pregnancy are recorded.

DETAILED DESCRIPTION:
Preterm birth is one of the leading causes for mortality and morbidity in newborns and preterm contractions are the cause of a considerable part of preterm deliveries. In the treatment of preterm labour, tocolytic medications are often used that are associated with numerous side effects for the pregnant woman, which limits their use in time. Preparations from Bryophyllum pinnatum, which demonstrated excellent tolerability, constitute a safe alternative for tocolytic treatment. It was introduced as an alternative tocolytic by anthroposophic medicine in Europe and is used as a monotherapy or add-on therapy for preterm labour in many perinatal clinics in Switzerland today. In vitro studies support the use of B. pinnatum as a tocolytic.

In addition, there are also limited options for the treatment of mental disorders and sleep disturbances during pregnancy. Anxiety plays a major role in the development of preterm labour and often leads to administration of tocolytics longer than necessary. Preparations from B. pinnatum have traditionally been in the treatment of anxiety. Improvements of sleep quality in pregnant women during treatment with B. pinnatum preparations were already shown in previous studies.

This exploratory study aims at investigating the effects of B. pinnatum for the treatment of anxiety in patients with signs of preterm birth.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Hospitalisation with signs of preterm birth
* Gestational age at randomisation >22 weeks (22+0) and <35 weeks (34+6)
* Good German or English skills
* Written informed consent

Exclusion Criteria:

* Early premature rupture of the membranes (PPROM)
* Factors that make soon delivery likely (pre-eclampsia, suspect cardiotocography, clinical signs of an amniotic infection)
* Body temperature >38°C
* Cervical opening or cervical length < 5 mm
* Contraindication for B. pinnatum, lactose or wheat protein allergy
* Taking Bryophyllum 50% chewable tablets or powder 48 h before study inclusion
* Taking psychotropic drugs (Benzodiazepines, antidepressants, neuroleptics)
* Diagnosed psychiatric disease (depression, anxiety disorder, adaptation disorder, post- traumatic stress disorder, bipolar disorder)
* Active participation in another interventional study during the last 4 weeks
* Known or suspected non-compliance with study protocol
* Drug or alcohol abuse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
change in situational state of anxiety | Assessment before treatment, after 1 week and after 2 weeks
  assessed with State-Trait-Anxiety-Inventory (STAI) values from 20 to 80, higher scores indicating worse state of anxiety
change in situational state of anxiety | assessment before treatment, after 1 week and after 2 weeks
  assessed with Pregnancy-related Anxiety Questionnaire Revised 2 (PRAQ-R2) values from 10 to 50, higher scores indicating worse state of anxiety

SECONDARY OUTCOMES:
change in sleep quality | assessment before treatment, after 1 week and after 2 weeks
  assessed with Pittsburgh Sleep Quality Index (PSQI) values from 0 to 21, higher scores indicating worse sleep quality
hospitalisation days | from randomisation till birth or end of preterm period, whichever came first, up to 9 weeks.
reached gestational age | at birth
incidence of Adverse Events | up to 9 weeks
  occurence of Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Background] Furer K, Simoes-Wust AP, von Mandach U, Hamburger M, Potterat O. Bryophyllum pinnatum and Related Species Used in Anthroposophic Medicine: Constituents, Pharmacological Activities, and Clinical Efficacy. Planta Med. 2016 Jul;82(11-12):930-41. doi: 10.1055/s-0042-106727. Epub 2016 May 24. PMID 27220081
- [Background] Plangger N, Rist L, Zimmermann R, von Mandach U. Intravenous tocolysis with Bryophyllum pinnatum is better tolerated than beta-agonist application. Eur J Obstet Gynecol Reprod Biol. 2006 Feb 1;124(2):168-72. doi: 10.1016/j.ejogrb.2005.05.013. Epub 2005 Jul 26. PMID 16051414
- [Background] Simoes-Wust AP, Jeschke E, Mennet M, Schnelle M, Matthes H, von Mandach U. Prescribing pattern of Bryophyllum preparations among a network of anthroposophic physicians. Forsch Komplementmed. 2012;19(6):293-301. doi: 10.1159/000345841. Epub 2012 Dec 17. PMID 23343584
- [Background] Lambrigger-Steiner C, Simoes-Wust AP, Kuck A, Furer K, Hamburger M, von Mandach U. Sleep quality in pregnancy during treatment with Bryophyllum pinnatum: an observational study. Phytomedicine. 2014 Apr 15;21(5):753-7. doi: 10.1016/j.phymed.2013.11.003. Epub 2013 Dec 25. PMID 24373544
- [Background] Simoes-Wust AP, Lapaire O, Hosli I, Wachter R, Furer K, Schnelle M, Mennet-von Eiff M, Seifert B, von Mandach U. Two Randomised Clinical Trials on the Use of Bryophyllum pinnatum in Preterm Labour: Results after Early Discontinuation. Complement Med Res. 2018;25(4):269-273. doi: 10.1159/000487431. Epub 2018 Jun 22. No abstract available. PMID 29945146
- [Background] Santos S, Haslinger C, Klaic K, Faleschini MT, Mennet M, Potterat O, von Mandach U, Hamburger M, Simoes-Wust AP. A Bufadienolide-Enriched Fraction of Bryophyllum pinnatum Inhibits Human Myometrial Contractility In Vitro. Planta Med. 2019 Mar;85(5):385-393. doi: 10.1055/a-0810-7704. Epub 2018 Dec 18. PMID 30562827
- [Background] Santos S, Haslinger C, Mennet M, von Mandach U, Hamburger M, Simoes-Wust AP. Bryophyllum pinnatum enhances the inhibitory effect of atosiban and nifedipine on human myometrial contractility: an in vitro study. BMC Complement Altern Med. 2019 Nov 4;19(1):292. doi: 10.1186/s12906-019-2711-5. PMID 31685022
- [Background] Santos S, Zurfluh L, Mennet M, Potterat O, von Mandach U, Hamburger M, Simoes-Wust AP. Bryophyllum pinnatum Compounds Inhibit Oxytocin-Induced Signaling Pathways in Human Myometrial Cells. Front Pharmacol. 2021 Feb 18;12:632986. doi: 10.3389/fphar.2021.632986. eCollection 2021. PMID 33679416